CLINICAL TRIAL: NCT00702949
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Evaluation of Pregabalin for Alleviating Hot Flashes
Brief Title: Pregabalin in Treating Women With Hot Flashes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N07C1; NCI-2012-02716 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000598191 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Pregabalin75 (Experimental): Patients receive 75 mg of oral pregabalin twice daily for 6 weeks.
  Interventions: Drug: pregabalin
- Pregabalin150 (Experimental): Patients receive 150 mg of oral pregabalin twice daily for 6 weeks.
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator): Patients receive oral placebo twice daily for 6 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: pregabalin — Given orally
  Arms: Pregabalin150; Pregabalin75
Other: placebo — Given orally
  Arms: Placebo

SUMMARY:
RATIONALE: Pregabalin may help relieve hot flashes in women with a history of breast cancer or those who have no history and do not wish to take estrogen therapy for fear of increased risk of breast cancer. It is not yet known what dose of pregabalin may be more effective in treating hot flashes.

PURPOSE: This is a randomized phase III trial to determine the efficacy of two doses of pregabalin, in comparison to placebo, in the prevention of hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of 150 mg of pregabalin versus placebo on hot flash scores in women with a history of breast cancer or women who do not wish to take estrogen therapy for fear of increased risk of breast cancer.
* To evaluate the side effect profile of different doses of pregabalin in these patients.
* To evaluate the effect of 150 mg of pregabalin versus placebo on the secondary outcome of interference of activities from hot flashes in these patients.
* To evaluate the efficacy and side effect profile of 75 mg of pregabalin versus placebo in these patients.

OUTLINE: Patients are stratified according to age (18-49 years vs ≥ 50 years); selective estrogen-receptor modulator (i.e., tamoxifen or raloxifene) or aromatase inhibitor use (yes vs no); duration of hot flashes (< 9 months vs ≥ 9 months); and frequency of hot flashes per 24-hour period (4-9 vs ≥ 10). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive 75 mg of oral pregabalin twice daily for 6 weeks.
* Arm II: Patients receive 150 mg of oral pregabalin twice daily for 6 weeks.
* Arm III: Patients receive oral placebo twice daily for 6 weeks. Treatment in all arms continues in the absence of unacceptable toxicity.

Patients complete Hot Flash Diaries at baseline and once daily during treatment and the Symptom Experience Diary at baseline and once weekly during treatment. Patients also complete the Profile of Mood States and the Hot Flash Related Daily Interference Scale questionnaires at baseline and after completion of study treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meeting 1 of the following criteria:

  * History of breast cancer (currently without malignant disease)
  * No history of breast cancer, but patient wishes to avoid estrogen due to a perceived increased risk of breast cancer
* Bothersome hot flashes (defined by their occurrence ≥ 28 times per week and of sufficient severity to make the patient desire therapeutic intervention)
* Presence of hot flashes for ≥ 1 month prior to study entry

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥ 6 months
* Able to complete questionnaire(s) by themselves or with assistance
* Women of childbearing potential not eligible (per the judgment of the attending clinician)
* Serum creatinine ≤ 1.5 times upper limit of normal

PRIOR CONCURRENT THERAPY:

* No prior gabapentin or pregabalin
* More than 4 weeks since prior and no concurrent antineoplastic chemotherapy, androgens, estrogens, or progestational agents

  * Vaginal estrogen is allowed if used for the past month and not planned to be discontinued
* Concurrent adjuvant targeted therapy (i.e., lapatinib, trastuzumab [Herceptin®]) allowed in patients with no evidence of disease
* Concurrent tamoxifen, raloxifene, or aromatase inhibitors on a constant dose for at least 4 weeks allowed provided the medication will not be stopped during the study period
* No concurrent or planned use of other agents for hot flashes except for any of the following:

  * Stable dose of vitamin E is allowed as long as agent was started > 30 days prior to study initiation and is to be continued throughout the study period
  * Soy is allowed, if it is planned to be continued at the same dose during the study period
  * Stable dose of antidepressants is allowed as long as it was started > 30 days prior to study initiation and is to be continued at a stable dose throughout the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, MD, Study Chair — Mayo Clinic
Locations (209):
- United States (209):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Loprinzi CL, Qin R, Stella PJ, et al.: Pregabalin for hot flashes in women: NCCTG trial N07C1. [Abstract] J Clin Oncol 27 (Suppl 15): A-9513, 2009.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 207 patients were enrolled on this trial between 06/20/2008, and 07/21/2008.
Pre-assignment Details: There were 16 cancels (6 in Arm I, 3 in Arm II and 7 in Arm III).
Period: Overall Study
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Started | 63 | 66 | 62
Evaluable for Primary Endpoint | 56 | 56 | 51
Completed | 58 | 57 | 54
Not Completed | 5 | 9 | 8
Not completed — Refusal | 3 | 2 | 2
Not completed — Adverse Event | 1 | 6 | 3
Not completed — Other Medical Reason/unknown | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo | Total
Number analyzed (Participants) | 63 | 66 | 62 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (10.6) | 60.6 (9.5) | 56.6 (6.4) | 60.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 62 | 191
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 66 | 62 | 191

OUTCOME MEASURES:

1. Primary Outcome: Numerical Change From Baseline in Hot Flash Score at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: Hot flash activity will be analyzed in a number of ways. For the primary analysis, the numerical change-from-baseline to hot flash score after week 6 of treatment will be compared between the highest dose treatment arm and the placebo arm. A hot flash score is computed for each patient by assigning points (1=mild, 2=moderate, 3=severe, 4=very severe) to each hot flash based on patient-reported severity, adding the points for each day, and averaging across each week of the study. Abbreviations for the analysis population description: Eligible patients (EPs). Evaluable for primary (EFP). Off-study for adverse event (AE). Do not have 6 weeks of data (NODATA).
Time Frame: Baseline, after week 6 of treatment
Population: Arm II: 66 EPs, 56 are EFP and 10 are not (2 off-study by refusal, 6 AE, 1 unknown reason and 1 NODATA). Arm III: 62 EPs, 51 are EFP and 11 are not (2 off-study by refusal, 3 AE, 3 NODATA and 3 due to other reasons).
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin150 | Placebo
Number analyzed (Participants) | 56 | 51
units on a scale | -9.6 [-12.9 to -7.6] | -6.1 [-7.9 to -2.9]
Statistical Analysis 1: Comparison: Pregabalin150 vs Placebo; Comparing the median numerical change from baseline on hot flash score for Pregabalin 150 Mg with the Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

2. Secondary Outcome: Numerical Change From Baseline in Hot Flash Frequency at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: The analysis of daily average hot flash frequency will follow as specified for the primary analysis. Abbreviations for the analysis population description: Eligible patients (EPs). Evaluable for primary (EFP). Off-study for adverse event (AE). Do not have 6 weeks of data (NODATA).
Time Frame: Baseline, after week 6 of treatment
Measure: Median (95% Confidence Interval); unit: Hot flashes per day
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Number analyzed (Participants) | 56 | 56 | 51
Hot flashes per day | -4.6 [-5.6 to -3.9] | -4.9 [-6.1 to -4.0] | -2.9 [-3.6 to -1.4]

3. Secondary Outcome: Percent Change From Baseline in Hot Flash Frequency at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: as for outcome 2
Time Frame: Baseline, after week 6 of treatment
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Number analyzed (Participants) | 56 | 56 | 51
percent change | -58.5 [-74.6 to -48.8] | -61.1 [-72.3 to -48.3] | -36.3 [-51.6 to -20.3]

4. Secondary Outcome: Comparison of 75 mg of Pregabalin vs Placebo, Numerical Change From Baseline in Hot Flash Score at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: Hot flash activity will be analyzed in a number of ways. For the this analysis, the numerical change-from-baseline to hot flash score after week 6 of treatment will be compared between the lower dose treatment arm and the placebo arm. A hot flash score is computed for each patient by assigning points (1=mild, 2=moderate, 3=severe, 4=very severe) to each hot flash based on patient-reported severity, adding the points for each day, and averaging across each week of the study. Abbreviations for the analysis population description: Eligible patients (EPs). Evaluable for primary (EFP). Off-study for adverse event (AE). Do not have 6 weeks of data (NODATA).
Time Frame: Baseline, after week 6 of treatment
Population: Arm I: 63 EPs, 56 are EFP and 7 are not (3 off-study by refusal, 1 AE, 2 NODATA and 1 due to other medical reasons). Arm III: 62 EPs, 51 are EFP and 11 are not (2 off-study by refusal, 3 AE, 3 NODATA and 3 due to other reasons).
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin75 | Placebo
Number analyzed (Participants) | 56 | 51
units on a scale | -9.7 [-12.1 to -7.3] | -6.1 [-7.9 to -2.9]
Statistical Analysis 1: Comparison: Pregabalin75 vs Placebo; Comparing the median numerical change from baseline on hot flash score for Pregabalin 75 Mg with the Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

5. Secondary Outcome: Comparison of 75 mg of Pregabalin vs Placebo. Percent Change From Baseline in Hot Flash Score at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: Hot flash activity will be analyzed in a number of ways. For the this analysis, the percent change-from-baseline to hot flash score after week 6 of treatment will be compared between the lower dose treatment arm and the placebo arm. A hot flash score is computed for each patient by assigning points (1=mild, 2=moderate, 3=severe, 4=very severe) to each hot flash based on patient-reported severity, adding the points for each day, and averaging across each week of the study. Abbreviations for the analysis population description: Eligible patients (EPs). Evaluable for primary (EFP). Off-study for adverse event (AE). Do not have 6 weeks of data (NODATA).
Time Frame: Baseline, after week 6 of treatment
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Pregabalin75 | Placebo
Number analyzed (Participants) | 56 | 51
percent change | -64.9 [-83.6 to -57.8] | -50.1 [-64.5 to -28.3]
Statistical Analysis 1: Comparison: Pregabalin75 vs Placebo; Comparing the median percent change from baseline on hot flash score for Pregabalin 75 Mg with the Placebo; Test type: Superiority or Other; p = 0.009, t-test, 2 sided

6. Secondary Outcome: Toxicity Data for the Individual Study Arms From the Symptom Experience Diary .
Description: A descriptive report of the toxicities experienced by participants will be measured with a Symptom Experience Diary. Participants will complete this questionnaire weekly. This patient diary contains several questions related to potential side effects and side benefits of pregabalin measured on a numeric analogue scale (based on 0-10 scale with 10 being worst toxicity, providing numbers representing the worst median changes from baseline minus Maximum (Week 1-6) Symptom Experience Diary Distributions).
Time Frame: Baseline, 6 weeks during treatment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Number analyzed (Participants) | 63 | 66 | 62
units on a scale
  Concern about weight gain | 1.0 [-2 to 10] | 2.0 [-2 to 10] | 1.0 [-9 to 10]
  Concern about sleepiness | 1.0 [-6 to 8] | 2.0 [-4 to 9] | 1.0 [-5 to 6]
  Concern about dizziness | 1.0 [-2 to 7] | 2.0 [-2 to 9] | 0 [-4 to 8]
  Concern about coordination | 0.0 [-3 to 6] | 1.0 [-3 to 9] | 0.0 [-3 to 8]
  Concern about concentration | 1.0 [-3 to 8] | 1.0 [-3 to 9] | 0.0 [-4 to 9]
  Concern about blurred/double vision | 0.0 [-3 to 7] | 1.0 [-1 to 7] | 0.0 [0 to 7]

7. Primary Outcome: Percent Change From Baseline in Hot Flash Score at Treatment Week 6 (Positive Numbers to Represent Increases and Negative Numbers to Represent Decreases).
Description: Hot flash activity will be analyzed in a number of ways. For the primary analysis, the percent change-from-baseline to hot flash score after week 6 of treatment will be compared between the highest dose treatment arm and the placebo arm. A hot flash score is computed for each patient by assigning points (1=mild, 2=moderate, 3=severe, 4=very severe) to each hot flash based on patient-reported severity, adding the points for each day, and averaging across each week of the study. Abbreviations for the analysis population description: Eligible patients (EPs). Evaluable for primary (EFP). Off-study for adverse event (AE). Do not have 6 weeks of data (NODATA).
Time Frame: Baseline, after week 6 of treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Pregabalin150 | Placebo
Number analyzed (Participants) | 56 | 51
percent change | -71.0 [-78.2 to -60.6] | -50.1 [-64.5 to -28.3]
Statistical Analysis 1: Comparison: Pregabalin150 vs Placebo; Comparing the median percent change from baseline on hot flash score for Pregabalin 150 Mg with the Placebo; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

8. Secondary Outcome: Mood and Hot Flash-related Daily Interference on Activities After 6 Weeks of Treatment
Description: Endpoints for this analysis will be median change from baseline to after week 6 of treatment. Hot Flash Related Daily Interference Scale is used to evaluate the specific impact of the study treatment on the effect hot flashes have on various life activities such as work, social, leisure and relationships. Responses to the questionnaire are recorded on a 0 to 10 scale. Lower scores are better.
Time Frame: Baseline, after week 6 of treatment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Number analyzed (Participants) | 63 | 66 | 62
units on a scale
  Work | -1.0 [-6 to 4] | -1.5 [-10 to 5] | -1 [-8 to 2]
  Social Activities | -1 [-7 to 4] | -1.5 [-8 to 4] | 0 [-7 to 7]
  Leisure Activities | -1 [-8 to 4] | -1 [-8 to 4] | 0 [-6 to 5]
  Sleep | -2 [-10 to 3] | -3 [-10 to 3] | -1 [-9 to 3]
  Mood | -1 [-7 to 4] | -1 [-8 to 6] | 0 [-7 to 7]
  Concentration | -1 [-7 to 6] | -1 [-7 to 4] | -1 [-8 to 5]
  Relations | -1 [-6 to 6] | 0 [-8 to 2] | 0 [-7 to 3]
  Sexuality | 0 [-5 to 4] | 0 [-9 to 2] | 0 [-9 to 7]
  Enjoy Life | -1 [-10 to 5] | -2 [-10 to 2] | -1 [-8 to 3]
  Overall QOL | -1.5 [-10 to 5] | -1.5 [-9 to 2] | 0 [-8 to 2]

ADVERSE EVENTS:
Arm/Group | Pregabalin75 | Pregabalin150 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/66 | 0/62
Other Adverse Events (participants affected / at risk) | 42/63 | 56/66 | 37/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin75 (N=63) | Pregabalin150 (N=66) | Placebo (N=62)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 3 (3) | 3 (4) | 0 (0)
Vision blurred (Eye disorders) | 10 (19) | 17 (25) | 9 (14)
Constipation (Gastrointestinal disorders) | 19 (38) | 28 (55) | 17 (33)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 13 (22) | 24 (40) | 16 (35)
Fatigue (General disorders) | 3 (5) | 3 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 11 (20) | 25 (41) | 11 (26)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 26 (48) | 35 (60) | 14 (28)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Orgasm abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes